CLINICAL TRIAL: NCT01966666
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential Cohort, Dose-Ranging Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of TPI-287 in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: A Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy Study of TPI-287 in Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Adam Boxer, Prinicpal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TPI287-AD-001
Record Dates: First submitted 2013-10-14; First posted 2013-10-21 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; mild to moderate
MeSH Terms: conditions — Alzheimer Disease | interventions — TPI-287

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TPI-287 low dose (Experimental): 2 mg/m2 of TPI-287 administered as a 1-hour intravenous infusion once every 3 weeks for 9 weeks (for a total of 4 infusions)
  Interventions: Drug: TPI-287 2 mg/m2; Drug: Placebo
- TPI-287 moderate dose (Experimental): 6.3 mg/m2 of TPI-287 administered as a 1-hour intravenous infusion once every 3 weeks for 9 weeks (for a total of 4 infusions)
  Interventions: Drug: TPI-287 6.3 mg/m2; Drug: Placebo
- TPI-287 high dose (Experimental): 20 mg/m2 of TPI-287 administered as a 1-hour intravenous infusion once every 3 weeks for 9 weeks (for a total of 4 infusions)
  Interventions: Drug: TPI-287 20 mg/m2; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TPI-287 2 mg/m2 — 2 mg/m2 of TPI-287 diluted with 500mL 0.9% sodium chloride. TPI-287 is a microtubule inhibitor belonging to the taxane diterpenoid (taxoid) family, and specifically to the abeotaxane class.
  Arms: TPI-287 low dose
Drug: TPI-287 6.3 mg/m2 — 6.3 mg/m2 of TPI-287 diluted with 500mL 0.9% sodium chloride. TPI-287 is a microtubule inhibitor belonging to the taxane diterpenoid (taxoid) family, and specifically to the abeotaxane class.
  Arms: TPI-287 moderate dose
Drug: TPI-287 20 mg/m2 — 20 mg/m2 of TPI-287 diluted with 500mL 0.9% sodium chloride. TPI-287 is a microtubule inhibitor belonging to the taxane diterpenoid (taxoid) family, and specifically to the abeotaxane class.
  Arms: TPI-287 high dose
Drug: Placebo — 500mL 0.9% sodium chloride.

SUMMARY:
The purpose of the study is to determine the highest dose of TPI-287 that is safe and tolerable when administered as an intravenous infusion to participants with mild to moderate Alzheimer's disease (AD), to measure pharmacokinetic properties of the drug as well as to gauge preliminary efficacy of TPI-287 on disease progression.

DETAILED DESCRIPTION:
The maximum tolerated dose of TPI-287 will be determined through a planned dose escalation over 3 sequential cohorts, each comprising of 11 participants randomized to either TPI-287 or placebo. TPI-287 or placebo will be administered as an intravenous infusion once every 3 weeks for 9 weeks, for a total of 4 infusions. Participants who successfully complete this phase will have the option of entering into the open label extension phase during which TPI-287 will be administered once every 3 weeks for an additional 6 weeks, for a total of 3 extra infusions.

Pre-medication of diphenhyramine 25 mg (Benadryl) will be given IV within 30 to 60 minutes prior to each study infusion in the study.

Safety and tolerability will be assessed through reporting of adverse events, physical and neurological testing, ECGs, as well as blood and urine analyses. Baseline and end-point measures of cognition and function, MRI brain scans, and cerebrospinal fluid (CSF) biomarker analyses will be used to determine preliminary efficacy of TPI-287 in mild-moderate AD. Pharmacokinetic and pharmacodynamic properties of TPI-287 will be calculated from blood plasma collected after the first infusion, and from CSF collected on the last visit of the placebo-controlled phase.

ELIGIBILITY:
Inclusion Criteria (all must be met):

1. Between 50 and 82 years of age (inclusive)
2. Meets National Institute on Aging-Alzheimer's Association Workgroups criteria for probable AD dementia (McKhann et al. 2011)
3. MRI at Screening is consistent with AD (≤ 4 microhemorrhages, and no large strokes or severe white matter disease)
4. MHIS at Screening is ≤ 4
5. MMSE at Screening is between 14 and 26 (inclusive)
6. FDA-approved AD medications are allowed as long as the dose is stable for 2 months prior to Screening. Other medications (except those listed under exclusion criteria) are allowed as long as the dose is stable for 30 days prior to Screening
7. Has a reliable study partner who agrees to accompany the subject to visits, and spends at least 5 hours per week with the subject
8. Agrees to 2 lumbar punctures
9. Signed and dated written informed consent obtained from the subject and the subject's caregiver in accordance with local IRB regulations
10. Males and all WCBP agree to abstain from sex or use an adequate method of contraception for the duration of the study and for 30 days after the last dose of study drug.

Exclusion Criteria (any one of the following will exclude a subject from being enrolled into the study):

1. Any medical condition other than AD that could account for cognitive deficits (e.g., active seizure disorder, stroke, vascular dementia)
2. History of significant cardiovascular, hematologic, renal, or hepatic disease (or laboratory evidence thereof)
3. History of significant peripheral neuropathy
4. History of major psychiatric illness or untreated depression
5. Neutrophil count <1,500/mm3, platelets <100,000/mm3, serum creatinine >1.5 x upper limit of normal (ULN), total bilirubin >1.5 x ULN, alanine aminotransferase (ALT) >3 x ULN, aspartate aminotransferase (AST) >3 x ULN, or INR >1.2 at Screening or baseline evaluations
6. Evidence of any clinically significant findings on Screening or baseline evaluations which, in the opinion of the Investigator would pose a safety risk or interfere with appropriate interpretation of study data
7. Current or recent history (within four weeks prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection
8. Current clinically significant viral infection
9. Major surgery within four weeks prior to Screening
10. Unable to tolerate MRI scan at Screening
11. Any contraindication to or unable to tolerate lumbar puncture at Screening, including use of anti-coagulant medications such as warfarin. Daily administration of 81 mg aspirin will be allowed as long as the dose is stable for 30 days prior to Screening
12. Subjects who, in the opinion of the Investigator, are unable or unlikely to comply with the dosing schedule or study evaluations
13. Any previous exposure to microtubule inhibitors (including TPI 287) within 5 years of Screening. Treatment with microtubule inhibitors other than TPI287 while on study will not be allowed
14. Participation in another AD clinical trial within 3 months of Screening
15. Treatment with another investigational drug within 30 days of Screening. Treatment with investigational drugs other than TPI 287 while on study will not be allowed
16. Known hypersensitivity to the inactive ingredients in the study drug
17. Pregnant or lactating
18. Positive pregnancy test at Screening or Baseline (Day 1)
19. Cancer within 5 years of Screening, except for non-metastatic skin cancer.

Ages: 50 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-11; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of TPI-287 | up to 13 weeks post initial dosing
  Planned dose range of intravenous infusions of TPI-287 administered once every 3 weeks for 9 weeks. The dose will be escalated in 3 sequential cohorts and participants will be monitored for adverse events to determine safety and tolerability.

SECONDARY OUTCOMES:
TPI-287 levels in blood plasma and cerebrospinal fluid | Screening and Week 10
  Blood plasma will be collected at specified time-points before and following the first infusion of study drug (TPI-287 or placebo) to measure TPI-287 levels. Steady-state levels of TPI-287 will be estimated from cerebrospinal fluid collected at end-point visit of placebo-controlled phase. These levels will be used to estimate the pharmacokinetic properties of TPI-287.

OTHER OUTCOMES:
CSF biomarkers of Alzheimer's disease | Screening and Week 10
  A lumbar puncture will be performed at the screening and final visits to obtain cerebrospinal fluid (CSF). CSF will be analyzed for changes to concentration of biomarkers of Alzheimer's disease - beta amyloid (1-42), total tau, phosphorylated tau, tau isoforms and fragments, and tau phosphopeptides.
Brain MRI scan | Screening and Week 11
  Brain MRI scans will be performed to explore effects of changes in brain network functional and structural connectivity as well as perfusion after administration of study drug.
Cognition | Screening and Week 11
  The Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-Cog) and Mini Mental State Examination (MMSE) will be conducted to determine effect and preliminary efficacy of the drug on cognition.
Degree of disability | Screening and Week 11
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) will be conducted to determine effect and preliminary efficacy of the drug on degree of disability.
Behavior | Screening and Week 11
  The Geriatric Depression Scale (GDS) will be conducted to determine effect and preliminary efficacy of the drug on behavior.
Number of participants with adverse events as a measure of safety and tolerability of extended administration of TPI-287 | up to 20 weeks post initial dosing
  Participants who successfully complete the placebo controlled phase will be offered the option to enter an open label extension phase comprising of 3 additional infusions of TPI-287, administered once every 3 weeks for 6 weeks. Participants will be monitored for adverse events to determine drug safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Adam L Boxer, M.D., Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Memory and Aging Center, San Francisco, California, United States

REFERENCES:
- [Derived] Tsai RM, Miller Z, Koestler M, Rojas JC, Ljubenkov PA, Rosen HJ, Rabinovici GD, Fagan AM, Cobigo Y, Brown JA, Jung JI, Hare E, Geldmacher DS, Natelson-Love M, McKinley EC, Luong PN, Chuu EL, Powers R, Mumford P, Wolf A, Wang P, Shamloo M, Miller BL, Roberson ED, Boxer AL. Reactions to Multiple Ascending Doses of the Microtubule Stabilizer TPI-287 in Patients With Alzheimer Disease, Progressive Supranuclear Palsy, and Corticobasal Syndrome: A Randomized Clinical Trial. JAMA Neurol. 2020 Feb 1;77(2):215-224. doi: 10.1001/jamaneurol.2019.3812. PMID 31710340